CLINICAL TRIAL: NCT00289159
Title: Follow Up by Multimodal MRI of a Cohort of Patients With Early Remitting Multiple Sclerosis (REPROMMS Study).
Brief Title: Multimodal MRI in Multiple Sclerosis (MS): Reliability and Follow Up
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Other Study IDs: RBM0110
Record Dates: First submitted 2006-02-08; First posted 2006-02-09 (Estimated); Last update posted 2006-02-09 (Estimated); Status verified 2005-09

CONDITIONS: Multiple Sclerosis
Keywords: aged 18-50; remitting evolution; less than two years of evolution; MS patients
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
To determine wether multimodal MRI (conventinal T1 and T2 sequences, diffusion, magnetization transfer, spectroscopy) is reproducible; to follow up a cohort of patients with early remmittent MS after treatment with interferon.

ELIGIBILITY:
Inclusion Criteria:

* MS patients according to Poser's criteria
* Remitting evolution (less than two years of evolution)
* Aged 18-50
* Immunomodulatory treatment indicated

Exclusion Criteria:

* Unable to perform MRI

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult

CONTACTS AND LOCATIONS:
Overall Officials: Ayman Tourbah, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris